CLINICAL TRIAL: NCT05223127
Title: Effect of Aloe Vera on Caesarean Section Wound Healing: Randomized Controlled Study
Brief Title: Aloe Vera on Caesarean Section Wound
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Hediye Karakoç, PhD Assistant Professor, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Karatay
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cesarean Section
Keywords: Aloe; Cesarean Section; Wound Healing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Aloe vera
  Interventions: Other: Aloe vera
- Control group (No Intervention): routine care (dressing with dry gauze)

INTERVENTIONS:
Other: Aloe vera — The leaves of Aloe vera (Aloe barbadensis) will be identified and verified by Selçuk University Faculty of Agriculture. Aloe vera leaves will be washed with antiseptic solution and cut crosswise using gloves and sterile knife. The thick epidermis will be removed from the middle of the leaf. The gel will be obtained from the parenchyma of the thick juicy leaves of aloe vera.
  Arms: Experimental group

SUMMARY:
Conducting clinical research in line with the literature recommendation, with a method that is low-cost, accessible, easy-to-use, and examined in an evidence-based design related to cesarean section wound, which negatively affects the quality of life of women in the postpartum period, constitutes the original value and our main motivation of the project.

DETAILED DESCRIPTION:
Cesarean section is the delivery of the fetus by incision in the abdominal and uterine wall and is a life-saving method when certain complications arise. While it was initially performed to take the baby alive from the mother who was about to die, it has become an easier operation with the developments in the field of surgery and anesthesia. In this direction, it has become a viable operation even at the request of the mother. However, there is no evidence of benefit to the mother or baby when applied when it is not necessary. In this direction, although the "ideal cesarean section rate" targeted by the World Health Organization since 1985 is between 10-15%, this rate is 37% in 2008, 48% in 2013 and 52% in 2018, according to Turkey Demographic and Health Research (TNSA) data. reported as. This situation brings many problems related to the postpartum period.

Cesarean section is a surgical intervention, not a form of delivery, and as with any surgical intervention, there are many risks. Moreover, the most important difference of cesarean section from any surgical intervention is that the fetus/newborn is also exposed to these risks. In addition, discomfort can be seen depending on the surgical procedure and the incision site after the cesarean section. In the study conducted to examine the cesarean section experiences and post-cesarean care needs of post-natal women; It is stated that almost all puerperant women have problems due to cesarean section, and pain is the leading problem, followed by pain, difficulty in movement, breastfeeding problem due to the incision site, gas, numbness and contraction while walking. It is stated that women who have had cesarean section most frequently experience problems related to their self-care in the early postpartum period, such as pain at the surgery site, difficulty in moving, gas formation, feeding and defecation. If these problems that occur in the mother during the postpartum period are not detected in a timely manner and are not intervened effectively, they can become chronic and negatively affect both the quality of life of the mothers and the health of the newborn.

Aloe vera is seen as an environmentally friendly traditional wound healing agent that increases collagen content and improves cross-links. It contains healing and moisturizing properties with its anti-inflammatory, antiviral, antibacterial, antifungal, antimicrobial properties. When the literature is examined, in the study on the use of aloe vera in cesarean wound healing; It is stated that no side effects of aloe vera gel were observed, the wound healing rate was higher in the first 24 hours in the intervention group, and there was no significant difference between the wound healing scores of the two groups at the end of the 8th day. However, it is recommended to conduct studies with longer interventions on the subject.

ELIGIBILITY:
Inclusion Criteria:

* In the age range of 18-35,
* Primiparous,
* Gestational week 37 and above,
* Transver incision made,
* Women who volunteered to participate in the study

Exclusion Criteria:

* Body mass index not in the range of 18.5-24.9,
* Having pregnancy complications (such as preeclampsia and diabetes),
* Having chronic diseases (such as anemia, coagulopathy, cardiovascular diseases and respiratory and kidney diseases),
* Smoking or substance use,
* Those who use drugs that affect wound healing (glucocorticoids, anticoagulants, immunosuppressants, antibiotics and chemotherapy drugs before cesarean section),
* Postpartum fever (≥38 ◦C),
* Conditions that cause excessive stretching of the uterus (multiple pregnancy, polyhydramnios),
* Self or baby in need of intensive care,
* Having had a hysterectomy or myomectomy during the operation,
* The operation takes more than 90 minutes,
* Individuals who do not want to withdraw from the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing | 12 hours
  It will be assessed using the REEDA scale.

SECONDARY OUTCOMES:
Ache | 12 hours
  It will be assessed using the McGill Pain Scale Short Form.
Life quality | 12 hours
  It will be assessed using the SF-36 Quality of Life Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hediye KARAKOC, PhD, Principal Investigator — KTO Karatay University

IPD SHARING:
Plan to Share IPD: No